CLINICAL TRIAL: NCT04631757
Title: A Prospective, Non-randomized, Phase II Study of Camrelizumab in Combination With Concurrent Chemoradiotherapy for Initial Unresectable Proximal Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma Conversion Therapy
Brief Title: Conversion Therapy of Camrelizumab Plus Chemoradiotherapy in Participants With Initial Unresectable Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-006
Record Dates: First submitted 2020-11-15; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus Chemoradiotherapy (Experimental): Patients with initial unresectable proximal gastric or gastroesophageal junction (GEJ) adenocarcinoma will receive camrelizumab 200mg q3w, SOX regimen (oxaliplatin 130mg/m2, d1, Q3w + S-1 40-60mg bid, d1-d14, Q3w), and intensity modulated radiotherapy for tumors and high-risk lymphatic drainage areas (45Gy/25d). Resectable patients after conversion therapy will receive D2 resection.
  Interventions: Drug: Camrelizumab + SOX + Radiotherapy

INTERVENTIONS:
Drug: Camrelizumab + SOX + Radiotherapy — Camrelizumab 200mg,d1,Q3w; oxaliplatin 130mg/m2, d1, Q3w; S-1 40-60mg bid, d1-d14,Q3w; intensity modulated radiotherapy 45Gy/25d

SUMMARY:
This is a study of Camrelizumab in Combination With concurrent radiotherapy and SOX for Initial Unresectable or potentially resectable proximal Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma. Patients without prior palliative therapy will be treated with Camrelizumab, radiotherapy (total 45 Gy), Oxaliplatin, and S-1. The primary endpoint is the 1-year PFS rate.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of Camrelizumab plus Concomitant Chemoradiotherapy in patients with Initial Unresectable or potentially resectable proximal Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma. 33 participants with Initial Unresectable locally advanced proximal gastric carcinoma /Gastroesophageal Junction (GEJ) Adenocarcinoma (Siewert type II/III) will be treated with conversion therapy as below once recruited:

1. induction chemotherapy (3w): one cycle of camrelizumab 200mg q3w and SOX regimen (oxaliplatin 130mg/m2, d1, Q3w + S-1 40-60mg bid, d1-d14,Q3w);
2. after the induction, concurrent Chemoradiotherapy will be started (5-6w): intensity modulated radiotherapy was given for tumors and high-risk lymphatic drainage areas, total dose:45Gy/25d, 1.8Gy/d, camrelizumab 200mg q3w, S-1 40-60mg bid, d1-d14, Q3w. The resectability assessment will be performed followed by MDT.
3. Participants still unresectable will receive additional conversion therapy with camrelizumab and SOX regimen. The resectability will be evaluated every 6 weeks until resectable or up to 8 cycles of conversion therapy.

Resectable patients will receive D2 resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provided written informed consent to be subjects in this trial.
* 18-75 years old.
* Has histologically-confirmed diagnosis of locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma.
* The initial unresectable or potentially resectable locally advanced proximal gastric carcinoma /Gastroesophageal Junction (GEJ) Adenocarcinoma (Siewert type II/III) in clinical stage T3-4N+M0 (AJCC 8 edition TNM stage) under any following condition: serious primary tumor invasion, unresectable bulky lymph node, retroperitoneal lymph node metastasis (RPLM). Clinical staging was performed according to enhanced CT/MRI examination.
* No prior systemic chemotherapy for the treatment of the participant's advanced or metastatic disease (include but not limited to surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy)
* Plan to have surgery after conversion therapy.
* Patients capable of taking oral medication.
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Survival expectation ≥12 months.
* Adequate organ function according to the following laboratory test results: absolute neutrophil count (ANC) ≥1.5×109/L; platelets ≥80×109/L; hemoglobin ≥90g/L; total bilirubin ≤1.5 ULN; serum creatinine ≤1.5 ULN or measured or calculated creatinine clearance > 50ml/min.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication and must be willing to use an adequate method of contraception for the course of the study through 90 days after the last dose of study medication. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy.

Exclusion Criteria:

* HER2 positive subjects will be excluded.
* With evidence of abdominal metastases.
* Has a known additional malignancy that is progressing within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
* The presence of any of the following cardiac clinical symptoms or diseases: New York Heart Association (NYHA) congestive heart failure of grade II or above, LVEF<50%, unstable angina pectoris, myocardial infarction within the past 12 months, QTc ≥ 450ms for male, QTc ≥ 450ms for female, electrocardiogram (ECG) examination revealed clinically significant abnormalities, have factors that increase the risk of prolonged QTc and abnormal heart rhythm.
* With active infection requiring drug intervention (e.g. anti-bacterial drugs, antiviral drugs, antifungal drugs treatment).
* Patients with active hepatitis B (HBsAg positive and HBV DNA≥500 IU/ml), hepatitis C (HCV antibodies positive and HCV RNA copies > ULN)
* With congenital immune deficiency or human immunodeficiency virus (HIV) infection.
* Plan to receive or have previously received an organ or allogeneic bone marrow transplant.
* Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, pulmonary function damaged seriously etc; active tuberculosis (TB).
* Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease.
* Who has received immunosuppressants/systemic corticosteroids therapy < 7 days before the first dose for an immunosuppression purpose (> 10mg/day prednisone or other equivalency drugs).
* Has received a live vaccine within 28 days prior to the first dose, plan to receive a live vaccine during or within 60 days after study treatment.
* Have any contraindications for study treatment.
* Participate in other clinical trials within 4 weeks before the first dose.
* Is pregnant or breastfeeding.
* Patients were judged unsuitable as subjects of this trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival (PFS) rate according to RECIST 1.1 base on investigator assessment | Up to approximately 12 months
  PFS was defined as the time from the first dose to the first documented disease progression per RECIST 1.1 based on investigator assessment. PFS rate at 1 year as estimated by Kaplan-Meier method.

SECONDARY OUTCOMES:
progression-free survival (PFS) according to RECIST 1.1 base on investigator assessment | Up to approximately 36 months
  PFS was defined as the time from the first dose to the first documented disease progression per RECIST 1.1 based on investigator assessment.
disease-free survival (DFS) Per RECIST 1.1 base on investigator assessment | Up to approximately 36 months
  DFS is defined as the time from post-surgery baseline scan until the first occurrence of local/distant recurrence or death from any cause and is based on RECIST 1.1 as assessed by investigators in patients undergoing surgery.
rate of R0-resections | Up to 30 days post-sugery
  the percentage of participants undergoing surgery with resection margin status negative.
Major pathological response（MPR） | Up to 30 days post-sugery
  The proportion of participants with a major pathological response (mPR) at the time of definitive surgery.
Pathological Complete Response (pCR) | Up to 30 days post-sugery
  Pathological complete response (pCR) is measured as the proportion of participants with a pathological complete response at the time of definitive surgery.
Overall Survival (OS) | Up to 5 years
  OS is the time from the first dose to death due to any cause.
Percentage of Participants Experiencing An Adverse Event (AEs) | Up to approximately12 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocolspecified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an adverse event. The number of participants who experienced an AE was reported for each arm according to the treatment received. The grade of AE will be assessed per CTCAE 5.0.